CLINICAL TRIAL: NCT02515708
Title: A Phase I Pilot Study to Assess Safety and Feasibility of Normothermic Machine Preservation In Human Liver Transplantation
Brief Title: Pilot Study to Assess Safety and Feasibility of Normothermic Machine Preservation In Human Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cristiano Quintini (Other)
Responsible Party: Sponsor-Investigator, Cristiano Quintini, Sponsor-Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-549
Record Dates: First submitted 2015-07-30; First posted 2015-08-05 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Normothermic Liver perfusion (Experimental): This group has the liver grafts preserved using the Normothermic Liver perfusion Device.
  Interventions: Device: Normothermic Liver perfusion Device
- Normothermic Machine Perfusion (single pump) (Other): This group has the liver grafts preserved using a single-pump variant of the Normothermic Liver perfusion Device.
  Interventions: Device: Normothermic Liver perfusion Device

INTERVENTIONS:
Device: Normothermic Liver perfusion Device — The liver grafts will be preserved at physiological temperature and have continuous perfusion with oxygen and nutrient supply in the ex vivo organ preservation phase.

SUMMARY:
Normothermic machine perfusion (NMP) preservation is a promising method to decrease the complication of marginal donor livers compared to cold storage (CS). The aim of this project is to assess safety and feasibility of NMP in human liver transplantation. This will be a single center prospective cohort pilot study. Thirty-two livers with acceptable quality for transplantation will be preserved with NMP in 2-18 hours and transplanted. The follow-up period will be 6 months post-transplantation. The outcome will be compared to 100 historical patients transplanted in our program in the past 5 years (liver preserved using CS) with matched characteristics on age, Model for End-Stage Liver Disease (MELD) score, preservation time, etc.

DETAILED DESCRIPTION:
The shortage of donor organs leads to the use of marginal donors including donors after cardiac death. Normothermic machine perfusion (NMP) preservation is a promising method to decrease their high risk of complication compared to the standard cold storage (CS). The aim of this project is to assess safety and feasibility of NMP in human liver transplantation.

This will be a single center prospective cohort pilot study. Thirty-two livers that have acceptable quality for transplantation will be preserved with NMP in 2-18 hours after cross clamp and cold flush. The liver grafts at NMP will be at physiological temperature and have oxygen and nutrient supply with continuous perfusion. The transplantation and post-transplant care will follow the standard of care. The follow-up period is 12 months after transplantation. The primary end point will be the rate of post-transplant Early Allograft Dysfunction (EAD), while the secondary end points will be: primary non function (PNF) rate, 1 and 6 months patient and graft survival, peak liver function tests in the first 7 days after transplantation, intraoperative hepatic arterial and portal flow measurement, rate and magnitude of post-reperfusion syndrome, surgical outcomes (operative time, transfusion requirement etc.), rate of post-transplant kidney failure, assessment of histological ischemia reperfusion (liver and bile duct), rate of vascular complications, rate of biliary complications, hospital and ICU length of stay, rejection rate, infection rate, the ability to predict function based on "on-pump" viability markers, and the incidence of adverse effect (AE).

The outcome will be compared to a control group of 100 historical patients (matched with a 1:4 ratio) transplanted in our program in the past 10 years (liver preserved using CS). Control subjects will be matched using donor and recipient age, Model for End-Stage Liver Disease (MELD) score, cold ischemia time, donor risk index and presence of steatosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary liver transplantation
* Age 18-75 years at the time of transplantation
* Willingness and ability to comply with the study procedures
* Signed Informed Consent Form
* For patients with hepatocellular carcinoma as indication for Orthoptic Liver Transplantation (OLT), tumor must be within Milan Criteria or down-staged to Milan Criteria.

Exclusion Criteria:

Recipient Exclusion Criteria:

* History of prior solid organ transplantation
* Patient on a respiratory and/or cardiocirculatory support at the time of transplant
* MELD score >35
* HIV positive patient
* Patient with current severe systemic infection
* Multiorgan transplant

Donor Exclusion Criteria:

* Donor age <14 or >70 years
* Liver steatosis (on visual estimate or on liver biopsy) > 30%
* Donors with Grade 2-3 traumatic liver laceration
* Partial grafts (living donors and split liver donors)
* Liver in which the investigator is unwilling or unable (for logistical reasons) to perform normothermic machine perfusion (NMP) preservation
* Inability to NMP perfuse the liver within 4 hours after cross clamp

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-05-16 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
the rate of Early Allograft Dysfunction post-transplantation in Normothermically Machine Perfused (NMP) livers | 7 days post-transplantation
  The presence of at least one of the following at post-transplant 7 days: serum bilirubin >= 10 mg/dL, international normalized ratio (INF) >= 1.6; and/or aspartate aminotransferase (AST) > 2000 U/L at any time in the first 7 post-transplant days (POD)

SECONDARY OUTCOMES:
primary non-function rate | in the first 10 days post-transplantation
graft survival | 6 months post-transplantation
  The allograft will be considered lost if a patient has a liver re-transplant or in the event of patient death.
peak liver function tests in the first 7 days post-transplantation | in the first 7 days post-transplantation
intraoperative flow measurement | intraoperative
  Flows will be measured with a transit time flowmeter (VeriQ system, MediStim A/S, Oslo, Norway) after graft reperfusion. The following parameters will be recorded as per our standard practice during liver transplantation: portal venous flow, hepatic artery flow, and hepatic artery flow after temporary portal vein occlusion.
post reperfusion syndrome (composite) | in the first 7 days post-transplantation
  rate and magnitude
surgical outcomes (composite) | intraoperative
  operative time, transfusion requirement
rate of post-transplant kidney failure | in the 1, 3, 6 ,9 months post-transplantation
histology of liver parenchyma | On the day of transplantation
vascular complications rate | in the first day post-transplantation
biliary complications rate | 6 months post-transplantation
hospital and ICU length of stay (composite) | 6 months post-transplantation
rejection rate | 6 months post-transplantation
opportunistic viral infection rate | 6 months post-transplantation
patient survival | 6 months post-transplantation
histology of bile duct | On the day of transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Cristiano Quintini, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No